CLINICAL TRIAL: NCT02708264
Title: Pessary in Prevention of Preterm Birth for Women With Twin Pregnancies and Short Cervical Length
Brief Title: Does Cervical Pessary Prevent Spontaneous Preterm Birth in Twin Pregnancies With Short Cervical Length?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Medical Doctor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 214/2015
Record Dates: First submitted 2016-03-06; First posted 2016-03-15 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcomes assessor and data analyst
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical Pessary (Experimental): The cervical pessary is a silicone device that has been used to prevent SPTB Pessary will be placed between 18 and 23 6/7 weeks gestation, and will be removed during the 36th week of pregnancy (or earlier if indicated)
  Interventions: Device: Cervical pessary
- No intervention (No Intervention): No pessary No pessary will be used. Subjects will receive standard obstetrical management

INTERVENTIONS:
Device: Cervical pessary — The cervical pessary is a silicone device that has been used to prevent SPTB
  Arms: Cervical Pessary

SUMMARY:
Spontaneous preterm birth (SPTB) remains the number one cause of perinatal mortality in many countries, including the United States. Multiple gestations are at increased risk of SPTB. A short cervical length (CL) on transvaginal ultrasound (TVU) has been shown to be a good predictor of SPTB, in both singletons and twins.

The cervical pessary is a silicone device that has been used to prevent SPTB. The efficacy of the cervical pessary has been assessed in several populations including singletons with short CL, unselected twins, twins with short CL, and triplet pregnancies. Several randomized clinical trials (RCTs) have been published, and several are ongoing. However, no consensus on use of the cervical pessary in pregnancy or guidelines for management have been assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Twin pregnancy (limits the participants to female gender)
* Short cervical length (less than or equal to 30 mm) on second trimester ultrasound at 18-23 6/7 weeks gestation

Exclusion Criteria:

* Singleton or higher order than twins multiple gestation
* Monoamniotic twins
* Twin twin transfusion syndrome
* Ruptured membranes
* Lethal fetal structural anomaly
* Fetal chromosomal abnormality
* Cerclage in place (or planned placement)
* Vaginal bleeding
* Suspicion of chorioamnionitis
* Ballooning of membranes outside the cervix into the vagina
* Painful regular uterine contractions
* Labor
* Placenta previa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Spontaneous Preterm delivery <34 weeks | Less than 34 weeks gestation

SECONDARY OUTCOMES:
Gestational age | Time of delivery
Birth weight | Time of delivery
Spontaneous preterm birth rates <37, <28 and <24 weeks | Less than 24, 28, 34 and 37 weeks gestation
Spontaneous rupture of membranes | Less than 34 weeks gestation
  Rupture of membranes <34 weeks
Type of delivery (if cesarean or operativa vaginal or spontaneous vaginal delivery) | Time of delivery
  cesarean delivery, operative vaginal delivery, spontaneous vaginal delivery
Neonatal death | Between birth and 28 days of age
Composite perinatal outcome | Between birth and 28 days of age
  Includes necrotizing enterocolitis, intraventricular hemorrhage (grade 3 or higher), respiratory distress syndrome, bronchopulmonary dysplasia (BPD), retinopathy, blood-culture proven sepsis and neonatal death
Maternal side effects | Maternal side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No